CLINICAL TRIAL: NCT01177306
Title: Phase 4 Study of the Effect of Extended Release Guanfacine on Working Memory in Children With ADHD
Brief Title: Inuniv and Working Memory
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lori A. Schweickert, MD (Individual)
Collaborators: Shire (Industry)
Responsible Party: Sponsor-Investigator, Lori A. Schweickert, MD, MD, Schweickert, Lori A., M.D.
Organization: Schweickert, Lori A., M.D. (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LAS-IST-001
Record Dates: First submitted 2010-07-29; First posted 2010-08-09 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD, working memory
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extended Release Guanfacine (Experimental): pre and post testing of working memory in subjects whose ADHD has responded to extended release guanfacine. Subjects will be tested before starting study drug and after 6-8 weeks on a stable dose of the study drug.
  Interventions: Drug: extended release guanfacine

INTERVENTIONS:
Drug: extended release guanfacine — 1-4 mg daily. Dose determined by response of ADHD symptoms to drug and by body mass limitations
  Other Names: Intuniv; Serial Number 306; IND 63,551

SUMMARY:
Minimum 24 subjects aged 8-12 with a diagnosis of ADHD will be prescribed extended release guanfacine (Intuniv) to assess impact, if any, on working memory. Pre and post testing using a standardized battery of tests for effect on symptoms of ADHD and working memory will be administered and assessed.

ELIGIBILITY:
Inclusion Criteria:

1.Meet DSM-IV criteria for ADHD, combined, inattentive, or hyperactive/impulsive subtype, as evidenced by minimum score of 24 on the ADHD-RS-IV at baseline

* 2 Outpatient status
* 3. Age 8-12 (inclusive) at baseline
* 4. Males or Pre-menarchal females
* 5. English-speaking parent and subject
* 6. If on stimulant medication, has demonstrated sub-optimal response to treatment ad is willing to be washed out (discontinued) from stimulant
* 7. Intellectual capacity to provide assent, as deemed by the Principal Investigator
* 8. No known cardiac history, including bradycardia, heart block, syncope or tachycardia
* 9. No known history of hypotension or hypotension at baseline
* 10. Willing to provide informed consent/ assent per IRB protocol

Exclusion Criteria:

* • 1.Meet DSM-IV criteria for ADHD, combined, inattentive, or hyperactive/impulsive subtype, as evidenced by minimum score of 24 on the ADHD-RS-IV at baseline

  * 2 Outpatient status
  * 3. Age 8-12 (inclusive) at baseline
  * 4. Males or Pre-menarchal females
  * 5. English-speaking parent and subject
  * 6. If on stimulant medication, has demonstrated sub-optimal response to treatment ad is willing to be washed out (discontinued) from stimulant
  * 7. Intellectual capacity to provide assent, as deemed by the Principal Investigator
  * 8. No known cardiac history, including bradycardia, heart block, syncope or or tachycardia
  * 9. No known history of hypotension or hypotension at baseline
  * 10. Willing to provide informed consent/ assent per IRB protocol 11. No history of hepatic or renal impairment

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Central Nervous System-Vital Signs (CNS-VS) | 6-8 weeks on stable dose of study drug
  standardized computer administered battery

SECONDARY OUTCOMES:
Wide Range Assessment of Memory and Learning(WRAML) | 6-8 weeks on stable dose of study drug
  psychologist administered battery assessing working memory

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Schweickert, MD, Principal Investigator — 3-C Family Services
Locations (1):
- 3C Family Services, Cary, North Carolina, United States

REFERENCES:
- [Result] Sallee FR, Lyne A, Wigal T, McGough JJ. Long-term safety and efficacy of guanfacine extended release in children and adolescents with attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2009 Jun;19(3):215-26. doi: 10.1089/cap.2008.0080. PMID 19519256
- [Result] Wang M, Ramos BP, Paspalas CD, Shu Y, Simen A, Duque A, Vijayraghavan S, Brennan A, Dudley A, Nou E, Mazer JA, McCormick DA, Arnsten AF. Alpha2A-adrenoceptors strengthen working memory networks by inhibiting cAMP-HCN channel signaling in prefrontal cortex. Cell. 2007 Apr 20;129(2):397-410. doi: 10.1016/j.cell.2007.03.015. PMID 17448997